CLINICAL TRIAL: NCT05013593
Title: The Effect of Red Clover Isoflavones on Urinary Microbiota Composition and Interaction With the Urothelium in Postmenopausal Women
Brief Title: Red Clover Isoflavones in Postmenopausal Women With Urge Urinary Incontinence and Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Annemarie Brusen Villadsen, Ph.D. student, Regionshospital Nordjylland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: N-20190028
Record Dates: First submitted 2021-08-03; First posted 2021-08-19 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Urge Incontinence; Overactive Bladder
Keywords: Microbiota; Microbiome
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo-controlled three-month trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Symptomatic RCE (Experimental): Bladder symptomatic group receiving red clover extract containing the two isoflavones formononetin and biochanin A. Isoflavone amount is 57.45 mg isoflavones daily (55.84 mg aglycones daily), in 70 ml red clover extract (35 ml twice daily, morning and evening with a meal)
  Interventions: Dietary Supplement: Red Clover Extract (RCE)
- Healthy RCE (Experimental): Healthy group without bladder symptoms receiving red clover extract containing the two isoflavones formononetin and biochanin A. Isoflavone amount is 57.45 mg isoflavones daily (55.84 mg aglycones daily), in 70 ml red clover extract (35 ml twice daily, morning and evening with a meal)
  Interventions: Dietary Supplement: Red Clover Extract (RCE)
- Symptomatic PL (Placebo Comparator): Bladder symptomatic group receiving placebo
  Interventions: Other: Placebo (PL)
- Healthy PL (Placebo Comparator): Healthy group without bladder symptoms receiving placebo
  Interventions: Other: Placebo (PL)

INTERVENTIONS:
Dietary Supplement: Red Clover Extract (RCE) — Red clover extract containing isoflavones Formononetin and biochanin A together with a heterogenous culture of probiotic lactic acid bacteria, and a natural sugar free raspberry/orange flavor. Isoflavone amount is 57.45 mg isoflavones daily (55.84 mg aglycones daily), in 70 ml red clover extract (35 ml twice daily, morning and evening together with a meal)
  Arms: Healthy RCE; Symptomatic RCE
Other: Placebo (PL) — Placebo containing water, brown coloring, and natural sugar free raspberry/orange flavor.
  Arms: Healthy PL; Symptomatic PL

SUMMARY:
The purpose of this study is to investigate the effect of red clover isoflavones in postmenopausal women with and without urge urinary incontinence and overactive bladder

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (more than 5 years since last menstruation)
* Read and understand Danish

Exclusion Criteria:

* Participants receive treatment with estrogen both oral, transdermal, and topical within three months prior to inclusion in the study
* Participants take estrogen-like compounds (isoflavones) three months prior to inclusion in the study
* Participants take prebiotic and/or probiotic supplements within three months prior to study inclusion
* Receive antibiotics (any) within three months prior to inclusion in the study
* Recurrent urinary tract infections (defined as ≥ 2 infections in the last six months or ≥ 3 infections during the last year)
* Acute urinary tract infection defined as positive urine culture and symptoms of acute cystitis
* Previous or current diseases of the digestive and/or urinary systems evaluated by PI (including, but not limited to inflammatory bowel disease (IBD) and cancer)
* Current or prior suffering from breast, ovary, and/or endometrial cancer
* Use hormone spiral within the last 5 years if they are under 60 years
* Hysterectomy before cessation of menstrual periods if the women are below the age of 60

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 108 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline microbiota composition in women suffering from UUI and OAB at three months follow-up | From baseline to three months follow-up
  The microbiota composition is analyzed using sequencing of bacterial DNA. We are investigating the urinary, vaginal and gut microbiota. In women with urge urinary incontinence (UUI) and overactive bladder (OAB) receiving RCE (symptomatic RCE), a possible change in the urinary, vaginal and fecal microbiota composition from baseline to three month follow-up, compared to controls receiving placebo (symptomatic PL) are investigated.
  Symptomatic RCE from baseline to follow-up vs. Symptomatic PL from baseline to follow-up
Change in baseline microbiota composition at three months follow-up | From baseline to three months follow-up
  The microbiota composition is analyzed using sequencing of bacterial DNA. Comparison of healthy women without bladder symptoms receiving RCE (healthy RCE) at baseline to three months follow-up compared to controls (healthy PL) from baseline to follow-up.
  Healthy RCE from baseline to follow-up vs. Healthy PL from baseline to follow-up
Difference in baseline microbiota composition between women with and without UUI and OAB | Baseline
  The microbiota composition is analyzed using sequencing of bacterial DNA. Is there a difference in the urinary, vaginal and gut microbiota in women with and without urge urinary incontinence (UUI) and overactive bladder (OAB) at baseline?
  Symptomatic PL baseline vs. Healthy PL baseline

SECONDARY OUTCOMES:
Comparison of the urinary, vaginal, and fecal microbiota | Baseline
  The microbiota composition is analyzed using sequencing of bacterial DNA. This composition is evaluated using alpha-diversity (measured based on number of unique bacteria as well as Shannon diversity and phylogenic diversity) and beta-diversity, as indicated by unifrac distance and bray-Curtis dissimilarity. Comparison of the urinary, vaginal, and fecal microbiota composition at baseline. All the different compartments are measured using the same Units of Measure.
  Healthy PL baseline urinary vs. Healthy PL baseline vaginal vs. Healthy PL baseline gut
Change in overactive bladder symptoms from baseline in women suffering from UUI and OAB at three months follow-up | From baseline to three months follow-up
  Overactive bladder symptoms are measured using the questionnaire International Consultation on Incontinence Questionnaire (ICIQ) Overactive Bladder (ICIQ-OAB). Comparison of symptom scores in women with UUI and OAB before and after treatment with RCE compared to placebo.
  Symptomatic RCE from baseline to follow-up vs. Symptomatic PL from baseline to follow-up
Change in urinary incontinence symptoms from baseline in women suffering from UUI and OAB at three months follow-up | From baseline to three months follow-up
  Urinary incontinence symptoms are measured using the questionnaire International Consultation on Incontinence Questionnaire (ICIQ) Urinary Incontinence Short Form (ICIQ-UI-SF). Comparison of symptom scores in women with UUI and OAB before and after treatment with RCE compared to placebo.
  Symptomatic RCE from baseline to follow-up vs. Symptomatic PL from baseline to follow-up
Change in blood estrogen levels from baseline to three months follow-up | From baseline to three months follow-up
  Blood estrogen levels are measured from serum blood samples. Blood samples are taken at baseline before RCE and PL intake and after three months treatment.
Change in blood isoflavone levels from baseline to three months follow-up | From baseline to three months follow-up
  Blood isoflavone levels are measured in ng/mL from plasma blood samples. Blood samples are taken at baseline before RCE and PL intake and after three months treatment.
Change in blood equol levels from baseline to three months follow-up | From baseline to three months follow-up
  Blood equol levels are measured in nmol/L from plasma blood samples. Blood samples are taken at baseline before RCE and PL intake and after three months treatment.
Change in gastrointestinal symptoms from baseline to three months follow-up | From baseline to three months follow-up
  Gastrointestinal symptoms are measured using Rom IV criteria before and after RCE and PL intake.
Change in Irritable Bowel Syndrome Severity Score Scale from baseline to three months follow-up | From baseline to three months follow-up
  Gastrointestinal symptoms are measured using the Irritable Bowel Syndrome Severity Score Scale before and after RCE and PL intake.
Change in Gastrointestinal Symptom Rating Scale from baseline to three months follow-up | From baseline to three months follow-up
  Gastrointestinal symptoms are measured using the Gastrointestinal Symptom Rating Scale before and after RCE and PL intake.

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie B Villadsen, Principal Investigator — Regionshospital Nordjylland
Locations (1):
- North Denmark Regional Hospital (Vendsyssel Hospital), Hjørring, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data will be shared upon article publication. Microbiome data (DNA sequences) will be uploaded to the Sequence Read Archive (SRA) at the National Center for Biotechnology Information (NCBI).
Time Frame: Data will become available upon article publication at NCBI.
Access Criteria: All will have access to the microbiome data